CLINICAL TRIAL: NCT01569581
Title: A Phase III Clinical Trial for Inactivated Enterovirus Type 71 Vaccine (Human Diploid Cell, KMB-17 Cell) in Chinese Infants and Children
Brief Title: A Protected Study of Inactivated EV71 Vaccine (Human Diploid Cell, KMB-17) in Chinese Infants and Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Medical Biology, Chinese Academy of Medical Sciences (Other)
Collaborators: Guangxi Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EV71-KMB17-III-IMB-CAMS
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: The Efficacy of Inactivated EV71 Vaccine (KMB17) Against HFMD in Chinese Children and Infants
Keywords: Human Enterovirus 71 (EV71); Hand, Foot and Mouth Disease (HFMD); Inactivated Vaccine; Human Diploid cell (KMB17); Adverse reactions associated with vaccine; Efficacy
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- 100U/0.5ml in 6-11 months old infants (Experimental): inactivated EV71 vaccine (KMB-17) of 100U/0.5ml (320Eu/0.5ml) in 1750 infants aged 6-11 months old on day 0, 28
  Interventions: Biological: 100U/0.5ml in 6-11 months old infants
- 100U/0.5ml in 12-23 months old infants (Experimental): inactivated EV71 vaccine (KMB-17) of 100U/0.5ml (320Eu/0.5ml) in 1750 infants aged 12-23 months old on day 0, 28
  Interventions: Biological: 100U/0.5ml in 12-23 months old infants
- 100U/0.5ml in 24-35 months old children (Experimental): inactivated EV71 vaccine (KMB-17) of 100U/0.5ml (320Eu/0.5ml) in 1500 children aged 24-35 months old on day 0, 28
  Interventions: Biological: 100U/0.5ml in 24-35 months old children
- 100U/0.5ml in 36-71 months old children (Experimental): inactivated EV71 vaccine (KMB-17) of 100U/0.5ml (320Eu/0.5ml) in 1000 children aged 36-71 months old on day 0, 28
  Interventions: Biological: 100U/0.5ml in 36-71 months old children
- 0U/0.5ml in infants (6-11 months old) (No Intervention): 0U/0.5ml (0Eu/0.5ml) placebo in 1750 infants aged 6-11 months old on day 0, 28
- 0U/0.5ml in infants (12-23 months old) (No Intervention): 0U/0.5ml (0Eu/0.5ml) placebo in 1750 infants aged 12-23 months old on day 0, 28
- 0U/0.5ml in children (24-35 months old) (No Intervention): 0U/0.5ml (0Eu/0.5ml) placebo in 1500 children aged 24-35 months old on day 0, 28
- 0U/0.5ml in children (36-71 months old) (No Intervention): 0U/0.5ml (0Eu/0.5ml) placebo in 1000 children aged 36-71 months old on day 0, 28

INTERVENTIONS:
Biological: 100U/0.5ml in 6-11 months old infants — inactivated EV71 vaccine (KMB-17) of 100U/0.5ml (320Eu/0.5ml) in 1750 infants aged 6-11 months old on day 0, 28
  Arms: 100U/0.5ml in 6-11 months old infants
Biological: 100U/0.5ml in 12-23 months old infants — inactivated EV71 vaccine (KMB-17) of 100U/0.5ml (320Eu/0.5ml) in 1750 infants aged 12-23 months old on day 0, 28
  Arms: 100U/0.5ml in 12-23 months old infants
Biological: 100U/0.5ml in 24-35 months old children — inactivated EV71 vaccine (KMB-17) of 100U/0.5ml (320Eu/0.5ml) in 1500 children aged 24-35 months old on day 0, 28
  Arms: 100U/0.5ml in 24-35 months old children
Biological: 100U/0.5ml in 36-71 months old children — inactivated EV71 vaccine (KMB-17) of 100U/0.5ml (320Eu/0.5ml) in 1000 children aged 36-71 months old on day 0, 28
  Arms: 100U/0.5ml in 36-71 months old children

SUMMARY:
Enterovirus 71 (EV71), a major pathogen that is responsible for causing hand-foot-and-mouth disease (HFMD) worldwide, is a member of the Human Enterovirus species A, family Picornaviridae.

Since the late 1990s, a series of large HFMD epidemics caused by EV71 have been reported in the Asia-Pacific region. Notably, there is evidence that the most severe cases from these epidemic outbreaks are associated with neurological disorders with CNS involvement caused by EV71 infection. Because of these EV71 infection-related public health issues, the research and development of EV71 vaccine candidates have been heavily promoted.

Recently, several EV71 vaccine candidates have been evaluated in animals but no final results of clinical trials, including inactivated vaccine, attenuated vaccine, subunit vaccine, DNA vaccine, epitope peptide vaccine, virus-like particles (VLPs).

Basing on the previous studies of elicited protection in mice and rhesus monkeys, a formalin-inactivated EV71 vaccine (Human Diploid cell, KMB-17 Cell) has been licensed by SFDA in China, Dec. 2010. The phase I clinical and phase II trials were completed, in Guangxi Province, China. The results of these clinical trials showed that this vaccine was safe and could induce effective antibodies for the infants. The purpose of phase III is to evaluate the protected and efficacy of the formalin-inactivated EV71 vaccine in Chinese infants and children (from 6 to 71 months old).

DETAILED DESCRIPTION:
Hand-foot-and-mouth disease (HFMD) is a significant cause of death, usually characterized by vesicular lesions on the skin and oral mucosa and high morbidity rates in children. Additionally, occasional fatal cases have been reported involving brainstem encephalitis and myelitis associated with cardiopulmonary collapse. Pulmonary edema/hemorrhage and respiratory failure are the major causes of death among children less than five years old.

Enterovirus 71 (EV71), a major pathogen that is responsible for causing HFMD worldwide, is a member of the Human Enterovirus species A, family Picornaviridae. Since the late 1990s, a series of large HFMD epidemics caused by EV71 have been reported in the Asia-Pacific region. Notably, there is evidence that the most severe cases from these epidemic outbreaks are associated with neurological disorders with CNS involvement caused by EV71 infection. Because of these EV71 infection-related public health issues, the research and development of EV71 vaccine candidates have been heavily promoted.

Recently, several EV71 vaccine candidates have been evaluated in animals but no final results of clinical trials, including heat-inactivated or formalin-inactivated vaccine, live-attenuated vaccine, recombinant viral protein 1 (VP1) vaccine, VP1 DNA vaccine, VP1 epitope peptide vaccine, EV71 virus-like particles (VLPs) and bacterial or viral vector expressing VP1. Overall, the inactivated whole-virus vaccines seem to be more immunogenic than recombinant VP1 and DNA vaccines.

Basing on the previous studies of elicited protection in mice and rhesus monkeys (Ying Zhang, et al. Pathogenesis study of Enterovirus 71 Infection in Rhesus Monkeys. Lab Invest, 2011, 91:1337-1350; Longding Liu, et al. Neonatal Rhesus Monkey is a Potential Animal Model for Studying Pathogenesis of EV71 Infection. Virology, 2011, 412:91-100; Chenghong Dong, et al. Immunoprotection Elicited by an Enterovirus Type 71 Experimental Inactivated Vaccine in Mice and Rhesus Monkeys. Vaccine, 2011, 29:6269-6275.), a formalin-inactivated EV71 vaccine (Human Diploid cell, KMB-17 Cell) has been licensed by SFDA in China, Dec. 2010. The phase I and phase II clinical trials were completed,in Guangxi Province, China.

The results showed that the formalin-inactivated EV71 vaccine (Human Diploid cell, KMB-17 Cell) was safety in Chinese adults (from 18 to 49 years old), children (from 3 to 11 years old) and infants (from 6 to 35 months old). This vaccine could induce specific cellular and humoral immune responses against EV71.

The phase III clinical trial will been carried out, from April 2012. The purpose of phase III is to evaluate the safety and efficacy of the formalin-inactivated EV71 vaccine in Chinese infants and children(from 6 to 71 months old) to protect them from EV71 infecting.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects (6-71 months infants) as established by medical history and clinical examination
* Full-term (37-42 weeks), weight ≥ 2500 g when it was born
* The subjects' legal guardian must be aware of this vaccines
* The subjects' legal guardian voluntarily participate in the study and signed Informed Consent Form
* Subjects with temperature ≤ 37.0℃
* The subjects' legal guardian with the ability and objective to comply with the requirements of the protocol
* Persist for a 2-month visit and receive blood tests according to program requirements

Exclusion Criteria:

* Subject who has a clinical diagnosis history of Hand, Foot and Mouth Disease (HFMD)
* Participated in the phase I or phase II clinical trails of the inactivated EV71 vaccine
* weight ≤ 2500 g when it was born
* Allergy or serious side-effects to a vaccine or any ingredient of vaccine
* Epilepsy, seizures, convulsions, neurological illness
* Congenital or hereditary immunodeficiency
* Autoimmune disease
* Severe malnutrition or dysgenopathy
* Asthma, thyroidectomy, angioneurotic edema, diabetes or cancer
* Asplenia, functional asplenia, and any circumstances leading to the asplenia or splenectomy
* Clinical diagnosis of coagulopathy (such as clotting factor deficiency, coagulation disorders, platelet abnormalities), significant bruising or blood clotting disorder
* Acute illness or acute exacerbation of chronic disease in last 7 days
* Any prior administration of immunodepressant or corticosteroids in last 6 months
* Any prior administration of blood products in last 3 months
* Any prior administration of live-attenuated vaccine in last 28 days or 1 months
* Any prior administration of subunit or inactivated vaccines in last 14 days Under the anti-TB prevention or therapy
* Fever before vaccination, axillary temperature ﹥37.0℃
* The laboratory test abnormalities before vaccination, including blood tests (hemoglobin, total white blood cells, WBC, platelets), blood biochemistry tests (ALT, total bilirubin, direct bilirubin, Cr, BUN) and urine tests (urine protein, urine sugar, blood cells), etc.
* Hypertension or hypotension. Systolic blood pressure ﹥140mmHg and/or diastolic blood pressure ﹥90mmHg; systolic blood pressure ﹤90mmHg and/or diastolic blood pressure ﹤60mmHg
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

Ages: 6 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12000 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of Inactivated EV 71 Vaccine (Human Diploid Cell, KMB-17) in Chinese Infants and children (from 6 to 71 months old) | within the first 28 days after the first vaccination
  Adverse reactions associated with vaccine and protection efficiency were observed in Chinese Infants and children (from 6 to 71 months old) after the first vaccination.
Evaluate the safety of Inactivated EV 71 Vaccine (Human Diploid Cell, KMB-17) in Chinese Infants and children (from 6 to 71 months old) | at the 28 days after the second vaccination
  Adverse reactions associated with vaccine were observed in Chinese Infants and children (from 6 to 71 months old) after the first vaccination.
Evaluate the efficacy of Inactivated EV 71 Vaccine (Human Diploid Cell, KMB-17) in Chinese Infants and children (from 6 to 71 months old) | within two years after the second vaccination
  The preventive efficacy were observed in Chinese Infants and children (from 6 to 71 months old) after the second vaccination

SECONDARY OUTCOMES:
Evaluate the seroconversion rate of anti-EV71 antibodies in serum of children and infant, after first vaccination | at the 28 day after the first vaccination
  The seroconversion rate of anti-EV71 antibodies was evaluated in serum of children and infant, at the 28 day after the first vaccination
Evaluate the seroconversion rate of anti-EV71 antibodies in serum of children and infant, after second vaccination | at the 28 days after the second vaccination
  The seroconversion rate of anti-EV71 antibodies was evaluated in serum of children and infant, at the 28 or 56 days after the second vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Zhaojun Mo, Master, Principal Investigator — Guangxi Provincial Center for Diseases Control and Prevention
Locations (1):
- Guangxi Provincial Center for Diseases Control and Prevention, Nanning, Guangxi, China

REFERENCES:
- [Derived] Zhang W, Kong Y, Jiang Z, Li C, Wang L, Xia J. Comprehensive safety assessment of a human inactivated diploid enterovirus 71 vaccine based on a phase III clinical trial. Hum Vaccin Immunother. 2016 Apr 2;12(4):922-30. doi: 10.1080/21645515.2015.1115934. Epub 2016 Feb 2. PMID 26837471
- [Derived] Liu L, Mo Z, Liang Z, Zhang Y, Li R, Ong KC, Wong KT, Yang E, Che Y, Wang J, Dong C, Feng M, Pu J, Wang L, Liao Y, Jiang L, Tan SH, David P, Huang T, Zhou Z, Wang X, Xia J, Guo L, Wang L, Xie Z, Cui W, Mao Q, Liang Y, Zhao H, Na R, Cui P, Shi H, Wang J, Li Q. Immunity and clinical efficacy of an inactivated enterovirus 71 vaccine in healthy Chinese children: a report of further observations. BMC Med. 2015 Sep 17;13:226. doi: 10.1186/s12916-015-0448-7. PMID 26381232
- [Derived] Li R, Liu L, Mo Z, Wang X, Xia J, Liang Z, Zhang Y, Li Y, Mao Q, Wang J, Jiang L, Dong C, Che Y, Huang T, Jiang Z, Xie Z, Wang L, Liao Y, Liang Y, Nong Y, Liu J, Zhao H, Na R, Guo L, Pu J, Yang E, Sun L, Cui P, Shi H, Wang J, Li Q. An inactivated enterovirus 71 vaccine in healthy children. N Engl J Med. 2014 Feb 27;370(9):829-37. doi: 10.1056/NEJMoa1303224. PMID 24571755